CLINICAL TRIAL: NCT02072746
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Effects of Daily Oral Zinc Sulfate (220 mg) in Subjects With Alcoholic Cirrhosis
Brief Title: Zinc Supplementation in Alcoholic Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Matthew Cave, Associate Professor, University of Louisville
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OICB10007; K23AA018399 (NIH)
Record Dates: First submitted 2014-02-19; First posted 2014-02-27 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Alcoholic Cirrhosis
Keywords: cirrhosis; alcohol
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Fibrosis | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc (Active Comparator): zinc sulfate 220 mg daily
  Interventions: Dietary Supplement: Zinc
- Placebo (Placebo Comparator): Placebo study for comparison
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc
  Other Names: Zinc sulfate 220 mg
  Arms: Zinc
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if zinc therapy: (1) strengthens your intestine's defensive barrier preventing damaging substances from reaching your liver, (2) decreases liver injury (inflammation, oxidative stress, cell death) and scarring, and (3) improves your liver-related health. Based on our preliminary animal data and other published reports, we expect zinc therapy to achieve all of these goals. Zinc is affordable, available over the counter or by prescription, and has an excellent safety profile. Positive results from this study will show that zinc is a significant therapy for millions of Americans with alcoholic liver disease.

DETAILED DESCRIPTION:
Two-thirds of Americans consume alcohol, and an estimated 14 million Americans are alcoholics. It has been estimated that 15%-30% of heavy drinkers develop advanced Alcoholic liver disease (ALD). The prevalence of ALD in the United States is conservatively estimated at 2 million persons. Nearly 50% of liver-related deaths and 30% of hepatocellular carcinomas in the US are due to alcoholic cirrhosis. Despite recent advances in our understanding of ALD, there is currently no FDA approved medication for any stage of ALD. Zinc sulfate is inexpensive, available over the counter, and has an excellent safety profile. If zinc positively influences the mechanisms postulated to play a role in human ALD, this affordable treatment would become relevant to millions of people worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Clinical diagnosis of alcoholic cirrhosis.
3. Between the ages of 18 years and 70 years.
4. Ability to attend all clinic visits and participate in monthly telephone calls.
5. Child-Pugh score of A or B.

Exclusion Criteria:

1. Allergy or intolerance to zinc sulfate.
2. Hospitalization within the previous 28 days.
3. Pregnancy.
4. Illicit drug use within the past 12 months.
5. Infection with hepatitis B, hepatitis C, or HIV.
6. Known or suspected cancer within the past 5 years.
7. Serum creatinine greater than 1.5 mg/dl within the past month.
8. Any severe chronic disease other than liver disease.
9. Impairment (slowness) of behavior, intelligence, and neuromuscular function which may indicate hepatic encephalopathy (slow or confused thinking due to your liver disease).
10. Participation in another clinical trial.
11. Any type of infection within the past month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Change in clinical status | Baseline to 3 months
  Whether the subject has improved clinically at time point.

SECONDARY OUTCOMES:
Blood zinc levels | 0,3,6,12,24 months
Change in serum endotoxin levels | 0,3,6,12,24 months
  Whether the subject has a change in the serum endotoxin levels.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cave, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States